CLINICAL TRIAL: NCT06950190
Title: Evaluating Cognitive Changes on Patients in Chemotherapy (ECCPC)
Acronym: (ECCPC)
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Ellis Medicine (Other)
Responsible Party: Principal Investigator, Dr.Tallat Mahmood,MD, Medical Oncologist, Ellis Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Chemotherapy-related Cognitive Impairment
Keywords: Cognitive Function; Cancer Survivorship; Cognitive Decline; Neurotoxicity; Chemotherapy; Chemobrain; Quality of Life; Behavioral Oncology
MeSH Terms: conditions — Chemotherapy-Related Cognitive Impairment; Cognitive Dysfunction; Neurotoxicity Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Intensity Walking Intervention (Experimental): Participants in this arm are asked to double their baseline daily step count ( which will be assessed for one week prior to start of chemo) using a pedometer. This low-intensity walking program is implemented alongside standard chemotherapy treatment with the aim of improving cognitive outcomes. Cognitive function is assessed using the MoCA at four time points (baseline and at three follow-up intervals during the study). Study staff provide regular monitoring and encouragement to help participants reach their step goals, making adjustments as needed to ensure safety and adherence.
  Interventions: Behavioral: Low-Intensity Walking Intervention
- Standard of Care (Control) (Other): Participants in this arm receive standard care during chemotherapy with no additional exercise intervention. They wear a pedometer for baseline step-count tracking but are not instructed to increase their activity beyond normal daily routines. This group serves as a comparison for the walking intervention group while maintaining usual activity levels. MoCA assessments are conducted at the same four scheduled time points (mirroring the experimental arm's schedule) to evaluate cognitive function without the influence of a prescribed exercise program.
  Interventions: Behavioral: Control Group Intervention

INTERVENTIONS:
Behavioral: Low-Intensity Walking Intervention — Participants in the experimental group will be asked to take part in a home-based, walking program. Each participant will receive a pedometer and will be instructed to increase their baseline daily step count by 100%. For example, if a participant typically walks 3,000 steps per day, they will be asked to increase their activity to 6,000 steps per day. Step counts will be regularly monitored, and participants will receive encouragement and support from study staff to help maintain adherence to the walking goals. In addition to the exercise intervention, participants in this group will undergo cognitive testing using the Montreal Cognitive Assessment (MoCA) at four timepoints: baseline, 6 months, 9 months, and 12 months. They will also complete self-reported questionnaires related to cognitive function at these same intervals. This group is designed to evaluate whether increased physical activity can improve or preserve cognitive function in patients undergoing chemotherapy.
  Arms: Low-Intensity Walking Intervention
Behavioral: Control Group Intervention — Participants in the control group will receive standard care and will not be given any specific exercise instructions. They will be provided with pedometers to track their daily steps, but they will not be asked to increase or change their usual level of physical activity. These participants will continue with their routine activities and cancer care as directed by their treating physicians. Like the intervention group, they will complete the Montreal Cognitive Assessment (MoCA) at baseline, 6 months, 9 months, and 12 months, as well as self-reported questionnaires about cognitive function at each timepoint. This group will serve as a comparator to determine the impact of the walking intervention on cognitive outcomes.
  Arms: Standard of Care (Control)

SUMMARY:
This randomized clinical trial aims to evaluate the impact of a structured low-intensity exercise program on cognitive function in adult cancer patients undergoing chemotherapy. The study enrolls 100 participants who are randomly assigned to either a standard care group or an exercise intervention group. Cognitive function is measured using the Montreal Cognitive Assessment (MoCA) at baseline, 6, 9, and 12 months. Participants in the intervention group are instructed to double their baseline daily step count, tracked via pedometer, while those in the control group maintain their usual activity. All patients are given the pedometer for one week prior to the start of chemo to monitor their step count and determine their baseline. The study also collects self-reported data on cognitive difficulties and psychological well-being. The primary objective is to determine whether regular physical activity mitigates chemotherapy-related cognitive decline ("chemo brain") and whether MoCA scores correlate with patients' subjective experiences. This low-cost, home-based approach may offer an accessible strategy for preserving cognitive function during cancer treatment.

DETAILED DESCRIPTION:
Chemotherapy-related cognitive impairment (CRCI) is a well-documented side effect of cancer treatment, yet its underlying mechanisms remain poorly understood and effective interventions are lacking. Emerging evidence suggests that physical activity may mitigate cognitive decline through improvements in neuroplasticity, cerebral blood flow, and reduction of inflammation-driven neurotoxicity. This study builds on that foundation by integrating both objective and subjective measures of cognitive function to better capture the patient experience. A mixed-effects ANCOVA model will be used to assess treatment effects over time, with additional analyses exploring the relationship between adherence to the exercise regimen and cognitive outcomes. By leveraging a low-cost, accessible intervention and including diverse demographic and psychosocial factors, this trial aims to inform future strategies for managing CRCI and improving long-term quality of life for cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* • Age 18 years and older.

  * Patients with histologically confirmed malignancy who are planning on receiving chemotherapy.
  * Able and willing to provide written informed consent.
  * ECOG performance status less than or equal to 2.
  * Patients willing and able to perform the exercise as directed.
  * Patients with the ability to walk without use of an assistive device.
  * Patients with no underlying psychiatric disorder (other than depression, as long as there has been no acute presentation within 6 months of being enrolled in the study).

Exclusion Criteria:

* • Under the age of 18 years.

  * Patients unable to provide informed consent.
  * Patients who are non-ambulatory or who have a physical disability preventing exercise.
  * ECOG performance status greater than 2.
  * Patients with a psychiatric diagnosis (other than depression)
  * Patients with a diagnosis of dementia of any type.
  * Patients with a neurologic disorder that one could reasonably assume to have an underlying cognitive impairment.
  * Patients with a history of traumatic brain injury.
  * Patients who will be on chemotherapy for longer than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2027-02-20 (Estimated); Study Completion 2027-02-20 (Estimated)

PRIMARY OUTCOMES:
Change in Cognitive Function as Measured by MoCA Score | Baseline, 6 months, 9 months, and 12 months
  This outcome evaluates whether cognitive decline associated with chemotherapy ("chemo brain") can be measured using the MoCA, a brief and validated tool suitable for clinical settings. The goal is to determine if MoCA can effectively detect changes in cognitive performance over the course of chemotherapy without the need for extensive neuropsychological testing.

SECONDARY OUTCOMES:
Correlation Between MoCA Scores and Self-Reported Cognitive Difficulties | Baseline, 6 months, 9 months, and 12 months
  This outcome examines how well participants' MoCA scores align with their own self-reported cognitive difficulties. Self-reported data will be collected using a structured questionnaire to capture subjective experiences of memory, attention, and mental clarity. The analysis will assess whether objective cognitive test results reflect participants' perceived impairments.

CONTACTS AND LOCATIONS:
Overall Officials: Tallat Mahmood, MD, Principal Investigator — Ellis Medicine/ Roswell Park
Locations (1):
- Ellis Medicine/Roswell Park Medical Oncology, Schenectady, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/23008308/
- See also: Related Info — https://www.cancer.org/research/cancer-facts-statistics/all-cancer-facts-figures/cancer-facts-figures-2022.html
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC4542053/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/28833160/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32091339/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/38552188/
- See also: Related Info — https://www.frontiersin.org/journals/psychology/articles/10.3389/fpsyg.2018.00509/full
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC5847033/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/20559064/
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC4842032/